CLINICAL TRIAL: NCT02366338
Title: PRescriptiOn PattERns Of Oral Anticoagulants in Non-valvular Atrial Fibrillation: A Single Center Experience From Turkey (PROPER)
Brief Title: PRescriptiOn PattERns Of Oral Anticoagulants
Acronym: PROPER
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ozcan Basaran, M.D., Muğla Sıtkı Koçman University
Other Study IDs: PROPER
Record Dates: First submitted 2015-02-08; First posted 2015-02-19 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial fibrillation is the major cause of acute ischemic stroke. The risk of stroke was shown to decline by oral anticoagulant therapy. The investigators intended to evaluate appropriate use of anticoagulants in non-valvular AF patients.

DETAILED DESCRIPTION:
Atrial fibrillation, the most common sustained arrhythmia, is the major cause of acute ischemic stroke. The prognosis of ischemic stroke associated with atrial fibrillation (AF) tends to have a worse prognosis for recovery compared with other ischemic stroke subtypes. The risk of stroke was shown to decline to 68% by oral anticoagulant (OAC) therapy.The investigators have evaluated appropriate use of anticoagulants in non-valvular AF patients. Appropriate use of oral anticoagulants was assessed by Medication Appropriateness Index (MAI). The MAI consists of 10 criteias namely, indication, choice, dosage, modalities and practicability of administration, drug-drug interactions, drug-disease interactions, duplication, duration, and cost-effectiveness. The tenth criteria was not evaluated because of limited data regarding cost-effectiveness of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Non valbular AF >18 years

Exclusion Criteria:

* Not currently receiving anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-valvular AF patients
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Basaran, Principal Investigator — Muğla Sıtkı Koçman University

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: patients on warfarin therapy
- Group 2: patients on rivaroxaban therapy
- Group 3: Patients on dabigatran therapy
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 73 | 39 | 36
Completed | 73 | 39 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 73 | 39 | 36 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9) | 69 (9) | 72 (8) | 71 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 22 | 20 | 84
  Male | 31 | 17 | 16 | 64
Region of Enrollment [Number; unit: participants]
  Turkey | 73 | 39 | 36 | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One Inappropriate MAI Criterion
Description: Appropriateness of oral anticoagulants was evaluated by adapted versions of the MAI
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 73 | 39 | 36
participants | 61 | 11 | 17

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 0/73 | 0/39 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No